CLINICAL TRIAL: NCT06709573
Title: Clinical Decision Support Assistance to Randomize Patients to Early or Late Adjunctive Vasopressin in Septic Shock
Brief Title: Early Versus Late Adjunctive Vasopressin in Septic Shock
Acronym: CASPER-Pilot
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Gretchen Sacha, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-547
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic Shock; Vasopressors; Vasopressin
MeSH Terms: conditions — Sepsis; Shock, Septic; Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early Vasopressin Initiation (Experimental): Patients randomized to this arm will have a provider BPA fire prompting vasopressin initiation when the norepinephrine dose is between 10-20 mcg/min
  Interventions: Drug: vasopressin - early initiation
- Standard of Care Vasopressin Initiation (Active Comparator): Patients randomized to this arm will have a provider BPA fire prompting vasopressin initiation when the norepinephrine dose is between 20-35 mcg/min
  Interventions: Drug: vasopressin - standard initiation

INTERVENTIONS:
Drug: vasopressin - early initiation — BPA fires to provider prompting vasopressin initiation when the norepinephrine dose is between 10-20 mcg/min
  Other Names: vasopressin
  Arms: Early Vasopressin Initiation
Drug: vasopressin - standard initiation — BPA fires to provider prompting vasopressin initiation when the norepinephrine dose is between 20-35 mcg/min
  Other Names: vasopressin
  Arms: Standard of Care Vasopressin Initiation

SUMMARY:
The goal of the CASPER-Pilot study is to develop clinical decision support (CDS) technology within Epic to randomize patients with septic shock to early versus standard of care vasopressin initiation. The primary aim of this study will be to test the hypothesis that CDS technology can be utilized to create two distinct cohorts of patients reflecting different times of vasopressin initiation based on norepinephrine dose requirements. Secondarily, this study will evaluate the proportion of patients whose norepinephrine dose at the time of vasopressin initiation is within the specified range for the intervention arm they were randomized to. Other outcomes of evaluation will include adherence to the developed CDS technology and comparison of clinical outcomes between the two treatment arms.

DETAILED DESCRIPTION:
Sepsis is a highly prevalent and morbid disease estimated to account for up to 20% of annual deaths globally. If not rapidly identified and intervened upon, patients with sepsis may progress to septic shock, which is associated with mortality rates up to 50%. Patients with septic shock have persistent hypotension requiring vasoactive agents to augment blood pressure despite fluid resuscitation. Norepinephrine is recommended first-line by the Surviving Sepsis Campaign (SSC) guidelines for patients with septic shock. If mean arterial pressure (MAP) remains inadequate on norepinephrine, vasopressin is suggested as the second-line adjunctive agent. Over 30% of patients with septic shock in the United States (US) receive adjunctive vasopressin, with use rising over time. Despite increased use over time, ideal patient selection and initiation timing for adjunctive vasopressin in the course of a patient's shock are not well elucidated. The 2021 iteration of the SSC guidelines note that initiating vasopressin when the patient requires between 0.25 and 0.5 mcg/kg/min of norepinephrine "seems sensible". Yet, many questions remain regarding the timing of vasopressin initiation. The goal of this proposal is to evaluate the timing of vasopressin initiation in patients with septic shock based on the norepinephrine requirements at the time of vasopressin initiation. This pilot study will attempt to develop CDS technology in which to answer this clinical question.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* Diagnosis of Septic Shock
* Admitted to Cleveland Clinic Main Campus Medical ICU
* Receiving continuous infusion of norepinephrine at a dose > 5 mcg/min at time of enrollment

Exclusion Criteria:

* Administration of any other vasoactive agent other than norepinephrine at time of enrollment
* Initiation of vasopressin by provider outside of the context of study when NE < 10 mcg/min (before BPA firing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Norepinephrine-equivalent dose | Outcome evaluated on day of vasopressin initiation
  The primary outcome is the norepinephrine-equivalent dose (in mcg/min) at the time of vasopressin initiation between patients who were randomized by CDS to early adjunctive vasopressin initiation compare to late adjunctive vasopressin initiation

SECONDARY OUTCOMES:
Proportion of patients within goal norepinephrine-equivalent dose range | Outcome evaluated on day of vasopressin initiation
  This outcome will evaluate the overall proportion of patients enrolled in the trial whose norepinephrine dose at the time of vasopressin is within the goal range for the treatment group (< 20 mcg/min for the early vasopressin group and > 20 mcg for the standard of care vasopressin)

OTHER OUTCOMES:
Hemodynamic Response | 6 hours after vasopressin initiation
  Compare rates of hemodynamic response to vasopressin initiation between patients who were randomized by CDS to early adjunctive vasopressin initiation compare to late adjunctive vasopressin initiation
ICU mortality | Through hospitalization admission
  Compare ICU mortality between patients who were randomized by CDS to early adjunctive vasopressin initiation compare to late adjunctive vasopressin initiation
In-hospital mortality | Through hospitalization admission
  Compare rates of in-hospital mortality between patients who were randomized by CDS to early adjunctive vasopressin initiation compare to late adjunctive vasopressin initiation
BPA response rates | between the time of study enrollment and vasopressin initiation
  Overall evaluate and describe BPA response: the proportion of patients who were initiated on vasopressin, time to vasopressin initiation after BPA firing, and provider documented rationale for not initiating vasopressin after BPA firing

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen L. Sacha, PharmD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacha GL, Lam SW, Wang L, Duggal A, Reddy AJ, Bauer SR. Association of Catecholamine Dose, Lactate, and Shock Duration at Vasopressin Initiation With Mortality in Patients With Septic Shock. Crit Care Med. 2022 Apr 1;50(4):614-623. doi: 10.1097/CCM.0000000000005317. PMID 34582425